CLINICAL TRIAL: NCT01869907
Title: Effect of Minocycline on Neuropathic Pain
Brief Title: Effect of Minocycline on Pain Caused by Nerve Damage
Acronym: EMON
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Pascal Vanelderen, Principal Investigator, Ziekenhuis Oost-Limburg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EMON
Record Dates: First submitted 2013-05-27; First posted 2013-06-05 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Neuropathic Pain Caused by Lumbar Radicular Pain
MeSH Terms: interventions — Minocycline; Amitriptyline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo, once daily
  Interventions: Drug: placebo
- Amitriptyline (Active Comparator): Amitriptyline 25mg, once daily
  Interventions: Drug: Amitriptyline
- Minocycline (Active Comparator): Minocycline 100mg, once daily
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline — 100 mg once daily by mouth during 14 days
  Arms: Minocycline
Drug: placebo — once daily by mouth during 14 days
  Arms: Placebo
Drug: Amitriptyline — 25mg once daily by mouth during 14 days
  Arms: Amitriptyline

SUMMARY:
The purpose of this study is to determine if minocycline is effective in the treatment of neuropathic pain. The effect of minocycline will be compared to the effect of placebo and amitriptyline.

DETAILED DESCRIPTION:
Neuropathic pain is pain caused by damage to the central or peripheral nervous system. To date, therapy consists of tricyclic antidepressants (such as amitriptyline) or anticonvulsants. However, results are disappointing. Minocycline, a FDA-approved second generation tetracycline, was efficacious in various animal models of neuropathic pain. We want to study the effect of minocycline in neuropathic pain in humans. The type of neuropathic pain we want to investigate is lumbar radicular pain since this is the most prevalent condition associated with neuropathic pain in humans.

This placebo-controlled randomized double blind trial consists of 3 arms:

1. Placebo, once daily by mouth during 14 days.
2. Amitriptyline 25mg, once daily by mouth during 14 days.
3. Minocycline 100mg, once daily by mouth during 14 days.

Patients can take rescue medication if necessary: tramadol 50mg by mouths up to 3-times daily.

Brain-derived neurotrophic factor is implicated in the generation and maintenance of neuropathic pain in different animal models of neuropathic pain. To study the role of brain-derived neurotrophic factor in neuropathic pain in humans, we will determine its concentration in serum and plasma before and after 14 days medication intake.

ELIGIBILITY:
Inclusion Criteria:

Lumbar radicular pain due to disc herniation, failed back surgery syndrome or spinal canal stenosis causing neuropathic pain

Exclusion Criteria:

1. Diabetic, alcoholic or drug induced polyneuropathies
2. Depression or psychiatric comorbidity affecting pain sensation.
3. Use of antidepressants
4. Fibromyalgia and Chronic Fatigue Syndrome
5. Pregnancy.
6. Previous spinal cord damage
7. Malignancies
8. Allergy to minocycline or amitriptyline

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Baseline (before start of study), 7 and 14 days after start of medication intake
  Pain intensity will be measured using a visual analogue scale and the change in pain intensity between baseline and day 7, day 7 and day 14, baseline and day 14 will be evaluated

SECONDARY OUTCOMES:
neuropathic pain diagnostic questionnaire (DN4) score | Baseline (before start of study), 7 and 14 days after medication intake
  The DN4 questionnaire is used to assess the neuropathic symptoms of the pain and the change in DN4 score between baseline and day 7, day 7 and day 14, baseline and day 14 will be evaluated
Amount of rescue medication taken | 7 and 14 days after medication intake
  Rescue medication consists of tramadol 50mg by mouth 3-times daily if necessary. Patients will be provided with a total of 42 tablets of tramadol 50mg for the duration of the study. The remaining rescue medication will be counted on day 7 and day 14 and the change in rescue medication intake between baseline and day 7, day 7 and day 14, baseline and day 14 will be evaluated

OTHER OUTCOMES:
Concentration of brain-derived neurotrophic factor (BDNF) in serum and plasma | Baseline (before start of study) and after 14 days of medication intake.
  A blood sample (10ml) will be taken at baseline and after 14 days medication intake. The concentration of brain derived neurotrophic factor will be determined by high sensitivity ELISA (R&D systems® Europe, United Kingdom; detection range: 20-4,000 pg/ml) and the change in BDNF-concentration in serum and plasma between baseline and day 14 will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Van Zundert, MD, PhD, Study Chair — Ziekenhuis Oost-Limburg; Martine Puylaert, MD, Study Chair — Ziekenhuis Oost-Limburg; Pieter De Vooght, MD, Study Chair — Ziekenhuis Oost-Limburg; Roel Mestrum, MD, Study Chair — Ziekenhuis Oost-Limburg; René Heylen, MD, PhD, Study Chair — Ziekenhuis Oost-Limburg; Pascal Vanelderen, MD, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

REFERENCES:
- [Result] Vanelderen P, Rouwette T, Kozicz T, Heylen R, Van Zundert J, Roubos EW, Vissers K. Effects of chronic administration of amitriptyline, gabapentin and minocycline on spinal brain-derived neurotrophic factor expression and neuropathic pain behavior in a rat chronic constriction injury model. Reg Anesth Pain Med. 2013 Mar-Apr;38(2):124-30. doi: 10.1097/AAP.0b013e31827d611b. PMID 23337936
- [Result] Bastos LF, de Oliveira AC, Watkins LR, Moraes MF, Coelho MM. Tetracyclines and pain. Naunyn Schmiedebergs Arch Pharmacol. 2012 Mar;385(3):225-41. doi: 10.1007/s00210-012-0727-1. Epub 2012 Jan 27. PMID 22282331
- [Result] Zhang Q, Peng L, Zhang D. Minocycline may attenuate postherpetic neuralgia. Med Hypotheses. 2009 Nov;73(5):744-5. doi: 10.1016/j.mehy.2009.04.028. Epub 2009 May 24. PMID 19467572
- [Result] Sumracki NM, Hutchinson MR, Gentgall M, Briggs N, Williams DB, Rolan P. The effects of pregabalin and the glial attenuator minocycline on the response to intradermal capsaicin in patients with unilateral sciatica. PLoS One. 2012;7(6):e38525. doi: 10.1371/journal.pone.0038525. Epub 2012 Jun 7. PMID 22685578